CLINICAL TRIAL: NCT03088800
Title: IBUPAP - Combination of Oral Ibuprofen and Acetaminophen (APAP) is Superior to Either Analgesic Alone for Pediatric Emergency Department (ED) Patients With Acute Pain
Brief Title: IBUPAP Study for Pain Management in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Co-Investigator, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-01-06
Record Dates: First submitted 2017-03-18; First posted 2017-03-23 (Actual); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-01

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oral Ibuprofen (Active Comparator): Oral Ibuprofen at 10mg/kg dose and placebo of equal volume
  Interventions: Drug: Ibuprofen
- Oral APAP (Active Comparator): Oral APAP at 15 mg/kg and placebo of equal volume
  Interventions: Drug: APAP
- Oral Ibuprofen and Oral APAP (Active Comparator): Oral Ibuprofen at 10mg/kg dose and APAP at 15mg/kg dose.
  Interventions: Drug: Ibuprofen; Drug: APAP

INTERVENTIONS:
Drug: Ibuprofen — Oral Ibuprofen at 10 mg/kg dose
  Arms: Oral Ibuprofen; Oral Ibuprofen and Oral APAP
Drug: APAP — Oral APAP at 15mg/kg dose
  Arms: Oral APAP; Oral Ibuprofen and Oral APAP

SUMMARY:
Current literature supports ibuprofen and APAP are the most commonly used analgesics in the pediatric ED for acute traumatic/non-traumatic pain. However, the analgesic benefits of combination ibuprofen and APAP in this specific setting does not exist, but instead only as it applies to pediatric patients with postoperative pain. Thus, we have designed a double-blind, randomized, controlled clinical trial to evaluate analgesic efficacy, safety and feasibility of combination therapy to potentially broaden its clinical application in the pediatric ED. The investigators' hypothesize that combination oral ibuprofen and APAP therapy is superior to either drug alone and is an excellent analgesic modality for controlling acute traumatic/non-traumatic pain in the pediatric ED.

DETAILED DESCRIPTION:
The investigators' hypothesize the combination of oral ibuprofen and acetaminophen (APAP) is superior to either analgesic alone plus placebo for pediatric emergency department patients with acute traumatic/non-traumatic pain

1. Intent to Treat, prospective, randomized, double-blind trial.
2. Primary outcome: Pain reduction via NRS/FACES pain scale at times 0 and 60 minutes from administration of medication(s).

   Secondary outcomes: Antipyretic effects, level of analgesia achieved with each patient diagnosis(es), incidence and type of adverse effect(s), and patients' and parents' satisfaction with achieved level of analgesia.
3. Population : ages 3 - 17. Sample size 90 patients (30 per arm). Group 1: oral ibuprofen at 10mg/kg dose and placebo of equal volume; Group 2: oral APAP at 15 mg/kg dose and placebo of equal volume; and, Group 3: oral ibuprofen at 10 mg/kg dose and APAP at 15mg/kg dose.
4. Location: Urban tertiary care hospital Pediatric ED with 40,000 annual departmental visits.
5. Duration of Enrollment: 1 year from commencement of the study.

6/7. Patients will be enrolled and randomized upon triage by an assigned nurse dedicated to the study into one of three groups by using a blocks-randomization scheme for every 15 patients maintained by the ED pharmacists.

8. For patients experiencing breakthrough pain, oral morphine sulfate at 0.2mg/kg will be provided.

Group 1: oral ibuprofen at 10 mg/kg dose and placebo of equal volume;

Group 2: oral APAP at 15 mg/kg dose and placebo of equal volume; and,

Group 3: oral ibuprofen at 10 mg/kg dose and APAP at 15mg/kg dose. Medications including placebo will be given via prefilled syringes of identical volume, color and flavor. Level of analgesia will be assessed at times 0 and 60 minutes from administration of medication(s).

All enrolled patients, health care practitioners, and research associates will be blinded to the study medication(s) given and to the allocation sequence. Pharmacist(s) who are aware of the study medication(s) will not enroll patients. The allocation sequence code will only be revealed to the researchers once recruitment, data collection, and data entry are completed.

ELIGIBILITY:
Inclusion Criteria:

* ages 3-17 years old presenting to the pediatric ED
* treating physician deems patient required ibuprofen Tylenol or both for pain relief

Exclusion Criteria:

* documented or suspected pregnancy, (2)
* parental refusal,
* allergies to NSAIDS or APAP
* inability to tolerate oral medications or contraindications to oral medication route
* received analgesics within 4 hours prior to ED presentation
* inability to use pain scales

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Motov, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Ibuprofen | Oral APAP | Oral Ibuprofen and Oral APAP
Started | 30 | 30 | 30
Completed | 30 | 30 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Ibuprofen | Oral APAP | Oral Ibuprofen and Oral APAP | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 30 | 90
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.20 (4.48) | 10.90 (3.98) | 12.17 (3.67) | 11.42 (4.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 10 | 33
  Male | 16 | 21 | 20 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 30 | 30 | 30 | 90
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Pain Score at 60 Minutes
Description: Pain Score via Numeric Rating Scale or FACES pain scale at 60 minutes from baseline ( ranging from 0 to 10, with 0 being no pain, 5 being moderate pain, and 10 being very severe pain)
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Ibuprofen | Oral APAP | Oral Ibuprofen and Oral APAP
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | 2.72 (2.15) | 3.10 (1.92) | 2.77 (2.08)

ADVERSE EVENTS:
Time Frame: 60 minutes
Arm/Group | Oral Ibuprofen | Oral APAP | Oral Ibuprofen and Oral APAP
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT03088800/Prot_SAP_000.pdf